CLINICAL TRIAL: NCT00077909
Title: Biomarkers and Protein Mass Expression Profiles in Bronchoalveolar Lavage From Patients With Lung Infiltrates
Brief Title: Study of Lung Proteins in Patients With Pneumonia
Status: Recruiting | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 040119; 04-CC-0119
Record Dates: First submitted 2004-02-12; First posted 2004-02-13 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-10-01

CONDITIONS: Pneumonia; Pulmonary Disease; Lung Disease
Keywords: Proteomics; Infection; Pneumonia; Mass Spectrometry; BAL; Natural History; Lung; Pulmonary Disease; Lung Infiltrates
MeSH Terms: conditions — Pneumonia; Lung Diseases; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patients with Infectious Pneumonia
- Group 2: Patients with Non-Infectious Pneumonia

SUMMARY:
This study will examine the different types of proteins present in the lungs of patients with pneumonia to explore the causes of different types of the disease. Pneumonia is a condition that causes lung inflammation AND is often caused by an infection. It is usually diagnosed by lung x-rays and listening to the chest with a stethoscope. This method can diagnose pneumonia, but it does not provide information on the cause of the inflammation - information that might be helpful in guiding treatment. This study will measure proteins in the lungs of patients to see if certain proteins are associated with specific forms of pneumonia, and can thus serve as biomarkers for disease.

Patients undergoing diagnostic bronchoscopy at the NIH Clinical Center may participate in this study. Patients will undergo bronchoscopy and bronchoalveolar lavage as scheduled for their medical care. For this procedure, the patient's mouth and throat are numbed with lidocaine; a sedative may be given for comfort. A thin flexible tube called a bronchoscope is advanced through the nose or mouth into the lung airways to examine the airways carefully. Saline (salt water) is then injected through the bronchoscope into the air passage, acting as a rinse. A sample of fluid is then withdrawn for microscopic examination. Researchers in the current study will use some of the fluid obtained from the lavage to examine for protein content.

In addition to the bronchoscopy and bronchoalveolar lavage, participants will have about 2 tablespoons of blood drawn to compare blood test results with the results of the lung washings. Patients' medical records will be reviewed to obtain information on past medical history, current medical treatment, vital signs, and results of x-ray tests.

DETAILED DESCRIPTION:
OBJECTIVE:

The objective of this study is to analyze bronchoalveolar lavage (BAL) fluid from patients with lung infiltrates in order to discover new biomarkers and protein/peptide expression patterns that are associated with specific types of pulmonary diseases and infections. Bronchoalveolar lavage (BAL) is a standard method to obtain lower airway samples to evaluate pulmonary infiltrates in order to diagnose infection, malignancy or non-infectious inflammation. After collecting the BAL (during a clinically indicated brochoscopy), samples are routinely sent to the clinical microbiology laboratory for stains, cultures and molecular analysis. We have recently developed a rapid, culture-independent method to identify unique peptide markers in BAL that identify specific bacterial species. We are expanding the scope of 04-CC-0119 that was based originally on collection of BAL supernatant only, to now collect, analyze and store whole (unprocessed) BAL. The availabilty of new methods of analyzing BAL will broaden the scope of the study to analyze BAL proteins, lung cells, and microbial pathogens. This will allow improved characterization of the host response to lung inflammation and infection and help to assess the feasibility of using the culture-independent approach on clinical BAL samples to identify specific pathogens.

POPULATION:

The study population will include all patients undergoing bronchoscopy for clinical indications at the Clinical Center who provide informed consent for chart review blood draw (optional), and analysis of BAL, as described in this protocol. We plan to acquire BAL samples that reflect a spectrum of community-acquired and opportunistic pathogens associated with pulmonary disease. In addition analysis of a range of non-infectious pulmonary processes (e.g. acute lung injury, acute respiratory distress syndrome and engraftment syndrome) is important to develop measures of sensitivity and specificity.

DESIGN:

This is a prospective observational study.

OUTCOME:

The expected outcome is to:

Develop a database of protein mass profiles of BAL fluid linked to specific microbiologic diagnoses.

To collect, analyze and store BAL to validate the usefulness of the genoproteomic culture-independent method of microbial identification.

To analyze lung cells associated with infectious or inflammatory pulmonary condidtions.

Our plan is to acquire 1,000 specimens from the Clinical Center with a range of clinical diagnoses including bacterial, viral, parasitic and fungal infections and sterile inflammation. When a sufficient number of samples in an individual category is collected (approximately 20-30), the samples will be analyzed with current proteomic techniques.

ELIGIBILITY:
* INCLUSION CRITERIA:
* All eligible patients undergoing diagnostic bronchoscopy who provide consent for proteomic analysis of BAL fluid supernatant and chart review of patient characteristics will be included in this study.
* A parent/guardian may provide consent for a child age 17 or under and a Legally Authorized Representative (LAR) may provide consent for adults unable to consent.

EXCLUSION CRITERIA:

Patients undergoing bronchoscopy but not wanting to participate with either the chart review or the proteomic analysis of BAL fluid supernatant will be excluded.

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient at the NIH Clinical Center who has a clinically indicated need for diagnostic bronchoscopy.@@@
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2004-02-20 (Actual)

PRIMARY OUTCOMES:
Peptide biomarker | Batch-driven analysis of samples.
  Detection of peptide biomarker for infectious disease as a cause of pneumonia.
Characterization of lung cells associated with pneumonia | Batch-driven analysis of samples.
  Analyze lung cells associated with infectious or inflammatory pulmonary conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony F Suffredini, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang H, Drake SK, Yong C, Gucek M, Lyes MA, Rosenberg AZ, Soderblom E, Arthur Moseley M, Dekker JP, Suffredini AF. A Genoproteomic Approach to Detect Peptide Markers of Bacterial Respiratory Pathogens. Clin Chem. 2017 Aug;63(8):1398-1408. doi: 10.1373/clinchem.2016.269647. Epub 2017 Jun 6. PMID 28588123
- [Background] Wang H, Drake SK, Yong C, Gucek M, Tropea M, Rosenberg AZ, Dekker JP, Suffredini AF. A Novel Peptidomic Approach to Strain Typing of Clinical Acinetobacter baumannii Isolates Using Mass Spectrometry. Clin Chem. 2016 Jun;62(6):866-75. doi: 10.1373/clinchem.2015.253468. Epub 2016 Apr 26. PMID 27117471
- [Background] Wang H, Drake SK, Youn JH, Rosenberg AZ, Chen Y, Gucek M, Suffredini AF, Dekker JP. Peptide Markers for Rapid Detection of KPC Carbapenemase by LC-MS/MS. Sci Rep. 2017 May 31;7(1):2531. doi: 10.1038/s41598-017-02749-2. PMID 28566732
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2004-CC-0119.html